CLINICAL TRIAL: NCT02613000
Title: Prospective, Multicenter Cohort Study on Prognostic Value of Gastrointestinal Symptoms and Intestinal-specific Biomarkers in Prediction of Outcome of Intensive Care Patients
Brief Title: Intestinal-Specific Organ Function Assessment (iSOFA Study)
Acronym: iSOFA
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Collaborators: Karolinska University Hospital (Other); Insel Gruppe AG, University Hospital Bern (Other); Vienna General Hospital (Other)
Responsible Party: Principal Investigator, Annika Reintam Blaser, Researcher, University of Tartu
Other Study IDs: iSOFA Study
Record Dates: First submitted 2015-11-18; First posted 2015-11-24 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Critical Illness; Multiple Organ Failure
MeSH Terms: conditions — Critical Illness; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In patients included in Part B, approx. 7 ml of arterial or venous blood will be drawn each morning during the study period. Standard EDTA containing vacutainers are used for blood sampling and placed into ice until centrifugation. Blood will be centrifuged at 4 degrees by study nurse or central laboratory of the study site, after which plasma will be separated and stored at -80 degrees in eppendorf vials containing 1 ml of plasma, marked and labelled with study code numbers.
  10 ml of urine will be sampled each morning Timing of admission day sample at time of plasma sampling (6 AM) from the collection bag and stored at -80 degrees. 2 eppendorf test-tubes containing 1 ml are used for urine sampling.
  Samples for citrulline measurements will be shipped to University of East Anglia, Norwich, United Kingdom and other samples to Maastricht University Medical Center, Netherland, for biochemical analyses to be performed.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- All enrolled patients/Group A: 500 consecutive adult patients will be enrolled in Part A (clinical data)
  Interventions: Other: No intervention
- Patients with blood and urine sampling/Group B: Patients with informed consent signed (anticipated 200 out of 500 patients) will participate in Part A (clinical data) and B (intestinal-specific biomarkers from blood and urine)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Importance of gastrointestinal (GI) function in critically ill patients has been recognized, but until now there is no validated clinical tool to monitor GI dysfunction as part of multiple organ dysfunction syndrome (MODS). The general aim of current project is to develop a five grade score (0-4 points) for assessment of GI function similar to SOFA sub-scores used for assessment of other organ systems. 500 consecutive adult patients admitted to the intensive care unit will be monitored for gastrointestinal symptoms, intra-abdominal pressure (IAP) and acute gastrointestinal injury (AGI) grades [1]. In 200 patients from these, plasma and urinary levels of possible biochemical markers of intestinal injury will be assessed.

Objectives:

* To determine the prognostic value of gastrointestinal symptoms alone and in combination with intra-abdominal pressure (IAP), and acute gastro-intestinal injury (AGI) grades in predicting the ICU-, 28 days and 90 days mortality of adult intensive care patients (Part A of the study)
* To describe the blood and urine levels of biochemical markers of intestinal injury in general cohort of intensive care patients (Part B of the study).
* To compare the prognostic values of the intestinal-specific plasma parameters (IFABP, citrulline, ILBP, and D-lactate) with the gastrointestinal symptoms, AGI grades, and the SOFA score in predicting of ICU-, 28 days and 90 days mortality of adult intensive care patients (Part B of the study) Study design: prospective, observational, multicenter study Patient population: All consecutive adult critically ill patients (25 to 50 patients for each study site, 500 patients in total) in need for intensive care admission during maximum 4 weeks of study period.

Duration of the study: for the individual patient 7 days and follow-up of 90 days Primary study outcome: 28 and 90 days all-cause mortality Secondary outcomes: ICU and hospital mortality, ICU length of stay, hospital length of stay, duration of mechanical ventilation, multiple organ failure as a cause of mortality, plasma and urinary levels of intestinal fatty-acid binding protein (I-FABP), citrulline, ileal lipid binding protein (ILBP), and D-lactate in general cohort of intensive care patients.

DETAILED DESCRIPTION:
Objectives

1. To determine the prognostic value of gastrointestinal symptoms alone and in combination with intra-abdominal pressure (IAP), and acute gastro-intestinal injury (AGI) grades in predicting the ICU-, 28 days and 90 days mortality of adult intensive care patients.
2. To describe the blood and urine levels of the intestinal-specific plasma parameters (I-FABP, citrulline, ILBP, and D-lactate) in general cohort of intensive care patients.
3. To compare the prognostic values of the intestinal-specific plasma parameters (I-FABP, citrulline, ILBP, and D-lactate) with the gastrointestinal symptoms, AGI grades, and the SOFA score in predicting of ICU-, 28 days and 90 days mortality of adult intensive care patients.

Hypothesis

1. GI symptoms, alone or in combination with IAP, and AGI grades as defined by WGAP statement improve the predictive capability of the SOFA score in critically ill patients.
2. Intestinal-specific plasma and urinary markers are good to excellent predictors of outcome in critically ill patients.
3. Best prediction is achieved by combination of GI symptoms, IAP and plasma markers.
4. A clinical score developed based on the data from this study can be combined with existing SOFA score and thereby the predictive value of the SOFA score will be improved.

To test these hypotheses, the study has two parts:

Part A. Clinical data and routine laboratory parameters of 500 consecutive patients will be collected for 7 days after ICU admission. Standard treatment is implemented; no additional interventions solely for the study will be performed. Waived consent is expected.

Part B. Blood and urinary samples for intestinal-specific laboratory markers will be drawn once daily from 200 patients enrolled in Part A, and analyzed in addition to standard clinical and laboratory data. First blood sample will be taken at admission to the intensive care unit. Informed consent will therefore be obtained from the patient or the next of kin after blood and urine sampling (delayed consent).

Research questions Part A.

1. What is the predictive capability of gastrointestinal symptoms, IAP and AGI grades in intensive care patients?
2. Does the use of the AGI grades or a new AGI score based on GI symptoms alone or in combination with IAP improve the predictive capability of the SOFA score in the intensive care patients? Part B.
3. What is the relationship between the intestinal-specific markers and the disease severity of the organ dysfunction, as described with the APACHE and the SOFA score?
4. What is the predictive value of the intestinal-specific markers in predicting ICU-, 28 days and 90 days all-cause mortality, ICU and hospital length of stay, and duration of mechanical ventilation?
5. Is there a correlation between the intestinal-specific markers and the gastrointestinal signs and symptoms?
6. Is the predictive value of the intestinal specific markers higher compared to the GI symptoms, IAP and AGI grades in predicting ICU-, 28 days and 90 days all-cause mortality, ICU and hospital length of stay, and duration of mechanical ventilation?
7. Does the addition of the intestinal-specific plasma and urinary markers increase the predictive value of the SOFA score in predicting outcome?
8. Is the combination of the intestinal-specific markers with the GI symptoms, IAP and AGI grades better in predicting outcome compared to two individual items?
9. What in these comparisons is the best marker or combination of markers?

Methods/design

1. Study design, setting and patient population This is a prospective multicenter cohort study where 500 consecutive adult patients admitted to the intensive care unit will be monitored for gastrointestinal symptoms, IAP and AGI grades. Of these 500 patients, 200 patients will be included in part B.

All consecutive adult critically ill patients (25 to 50 patients for each study site) in need for intensive care admission during maximum 6 weeks.

The study will consist of three phases:

1. Screening assessment, documentation of admission parameters;
2. Study period of 7 days for the individual patient;
3. Follow-up period of 90 days.

2. Study sites and the duration of the study The study will be conducted in ICUs of both university teaching hospitals and general (non-academic) hospitals. 20 ICUs from different countries will be invited and expected to participate, and each site is expected to enrol 25 to 50 patients during the maximum period of 6 weeks.

For individual patient the study period is 7 days or till ICU discharge and follow-up of 90 days.

ELIGIBILITY:
Part A Inclusion criteria

* Admission to ICU during the study period (the patients already in the ICU at the time the study starts will not be included)
* Age at least 18 years Exclusion criteria
* Age <18 years
* Restriction of care at admission (i.e any limitation of intensive care measures)
* Readmission 7 or more days after initial admission to ICU

Part B Inclusion criteria

* Admission to ICU during the study period (the patients already in the ICU at the time the study starts will not be included)
* Age at least 18 years
* Signed informed consent by patient or next of kin or legal representative for blood sampling.

Exclusion criteria

* Age <18 years
* Restriction of care at admission (i.e any limitation of intensive care measures)
* Readmission 7 or more days after initial admission to ICU
* Absence of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult critically ill patients (25 to 50 patients for each study site, 500 patients in total) in need for intensive care admission during maximum 6 weeks of study period.
Sampling Method: Non-Probability Sample
Enrollment: 544 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tartu University Hospital, Tartu, Estonia

REFERENCES:
- [Derived] Padar M, Starkopf J, Starkopf L, Forbes A, Hiesmayr M, Jakob SM, Rooijackers O, Wernerman J, Ojavee SE, Reintam Blaser A. Enteral nutrition and dynamics of citrulline and intestinal fatty acid-binding protein in adult ICU patients. Clin Nutr ESPEN. 2021 Oct;45:322-332. doi: 10.1016/j.clnesp.2021.07.026. Epub 2021 Aug 3. PMID 34620335
- [Derived] Reintam Blaser A, Padar M, Mandul M, Elke G, Engel C, Fischer K, Giabicani M, Gold T, Hess B, Hiesmayr M, Jakob SM, Loudet CI, Meesters DM, Mongkolpun W, Paugam-Burtz C, Poeze M, Preiser JC, Renberg M, Rooijackers O, Tamme K, Wernerman J, Starkopf J. Development of the Gastrointestinal Dysfunction Score (GIDS) for critically ill patients - A prospective multicenter observational study (iSOFA study). Clin Nutr. 2021 Aug;40(8):4932-4940. doi: 10.1016/j.clnu.2021.07.015. Epub 2021 Jul 18. PMID 34358839